CLINICAL TRIAL: NCT04387942
Title: The Therapeutic Value and Mechanism of Recombinant Human Interleukin-2 in Children With Henoch-schönlein Purpura
Acronym: HSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20K012-001
Record Dates: First submitted 2020-05-06; First posted 2020-05-14 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Purpura, Schoenlein-Henoch
Keywords: HSP
MeSH Terms: conditions — IgA Vasculitis | interventions — Interleukin-2; aldesleukin; Injections

STUDY DESIGN:
Intervention Model Description: group A:patients were treated with IL-2.group B:patients were not treated with IL-2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Interleukin-2 (Experimental): patients were treated with IL-2.
  Interventions: Drug: IL-2
- Traditional therapy (No Intervention): patients were treated with dipyridamole and/or glucocorticoid，immunosuppressor.

INTERVENTIONS:
Drug: IL-2 — For all patients,rhIL-2 infusions seven days;recurrent patients was applied again for 7 days;patients who were diagnosed HSPN were treated on a routine basis for 7 consecutive days, and then once every two week for 3months.
  Other Names: Recombinant Human Interleukin-2 for Injection
  Arms: Recombinant Human Interleukin-2

SUMMARY:
The study aims to explore the therapeutic value and mechanism of Interleukin-2 on children with Henoch-schönlein purpura.

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study that routinely administered low-dose IL-2 therapy to monitor the improvement of clinical and laboratory parameters to explore its efficacy and to observe changes in immune cell subsets and cytokines.For all patients,rhIL-2(500,000 unit per square meter) infusions seven days;recurrent patients were applied again for 7 days;patients who were diagnosed HSPN were treated on a routine basis for 7 consecutive days, and then once every two week for 3months.

ELIGIBILITY:
Inclusion Criteria:

1. age <18 years old
2. meet the EULAR/PRINTO/PRES for the diagnosis of HSP
3. HIV negative;Negative for HBV and HCV.

Exclusion Criteria:

1. heart failure (cardiac function ≥ grade III NYHA)
2. liver insufficiency (upper limit of normal range of transaminase > 2 times)
3. renal insufficiency (creatinine clearance ≤30ml/min)
4. acute or severe infections such as bacteremia and sepsis
5. malignant tumor
6. high-dose steroid pulse therapy or intravenous injection of glucocorticoids in the last 1 month
7. mental disorders or any other chronic illness or substance abuse may interfere with the ability to comply with agreements or provide information
8. Intestinal ischemia or perforated gastrointestinal bleeding requires surgery
9. Inability to comply with IL-2 treatment regimen.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The change of immunological responses | day 0,day 7
  Enumeration of the number of subjects with a change in the absolute number of immune cells and serum cytokines in the peripheral blood

SECONDARY OUTCOMES:
The value of serum immunoglobulins and complements | day 0,day 7,3 month,6 month
  Laboratory measures were detected, including,serum total IgE, serum Ig A,serum IgG,serum IgM,C3 and C4.
Incidence of adverse drug reactions | up to 6 month
  Adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor, cardiovascular event,drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Yang si rui, MD and PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Sirui Yang, Changchun, Changchun/JiLin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St John J, Vedak P, Garza-Mayers AC, Hoang MP, Nigwekar SU, Kroshinsky D. Location of skin lesions in Henoch-Schonlein purpura and its association with significant renal involvement. J Am Acad Dermatol. 2018 Jan;78(1):115-120. doi: 10.1016/j.jaad.2017.04.1122. PMID 29241772
- [Background] Jen HY, Chuang YH, Lin SC, Chiang BL, Yang YH. Increased serum interleukin-17 and peripheral Th17 cells in children with acute Henoch-Schonlein purpura. Pediatr Allergy Immunol. 2011 Dec;22(8):862-8. doi: 10.1111/j.1399-3038.2011.01198.x. Epub 2011 Sep 19. PMID 21929599
- [Background] Fontenot JD, Rasmussen JP, Gavin MA, Rudensky AY. A function for interleukin 2 in Foxp3-expressing regulatory T cells. Nat Immunol. 2005 Nov;6(11):1142-51. doi: 10.1038/ni1263. Epub 2005 Oct 16. PMID 16227984
- [Background] Ross SH, Cantrell DA. Signaling and Function of Interleukin-2 in T Lymphocytes. Annu Rev Immunol. 2018 Apr 26;36:411-433. doi: 10.1146/annurev-immunol-042617-053352. PMID 29677473